CLINICAL TRIAL: NCT03145740
Title: The Effect of Intensive Facial Oral Tract Therapy (F.O.T.T.®) on Swallowing Function in Patients After Acquired Brain Injury (ABI)
Brief Title: Intensive Faciltiation of Swallowing in Patients With Severe Dysphagia After Acquired Brain Injury
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rigshospitalet, Denmark (Other)
Collaborators: Unfallkrankenhaus Berlin (Other)
Responsible Party: Principal Investigator, Ingrid Poulsen, Head of Research Unit, Rigshospitalet, Denmark
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: H-2-2013-162
Record Dates: First submitted 2017-04-10; First posted 2017-05-09 (Actual); Last update posted 2017-05-09 (Actual); Status verified 2017-05

CONDITIONS: Deglutition Disorders
MeSH Terms: conditions — Deglutition Disorders

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: The patient´s primary physician in the clinic, the primary occupational therapist, physiotherapist and the nurses were kept blinded for the whole period of the intervention.
  The patient´s relatives did know into what group the patient was randomized. The patient himself did not know. The occupational therapists associated to the project were not blinded.
  The otolaryngologist, who scored the video recorded FEES examinations was blinded. The colleagues from Germany, who analyse data are blinded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intensive F.O.T.T.® (Experimental): Intensive F.O.T.T.® intervention was given twice a day, approximately 20 minutes per intervention, exclusive time to position the patient. Before and after the intervention, the patient was positioned in a standardized way in side lying for 10 minutes to rest. Here, the Electromyographic Bioimpedance Measuring device (EMBI) measured the spontaneous swallowing frequency and -quality during both, the resting period and the intervention. In the intervention itself, the patient was facilitated with specific handling and interventions to swallow, according to F.O.T.T.®. The faciltation was embedded into a meaningful context for the patient, e.g. tooth brushing or eating small amounts of apple sauce, if safe.
  Interventions: Other: Intensive F.O.T.T.®
- Unspecific stimulation of face and mouth (Placebo Comparator): The intervention in the control group was given twice a day, approximately 20 minutes per intervention, exclusive time to position the patient. Patients in the control group were before and after the intervention, positioned in a standardized way in side lying for 10 minutes to rest. The EMBI measured the spontaneous swallowing frequency and -quality during both, the resting period and the intervention. The intervention included unspecific stimulation of the hands and the face, without therapeutic interventions directed towards facilitation of swallowing.
  Interventions: Other: Unspecific Stimulation of face and mouth

INTERVENTIONS:
Other: Intensive F.O.T.T.® — Therapeutic F.O.T.T.® intervention provided by Occupational Therapists (OTs). The intervention consists of positioning the patient, and giving sensory input to the hands and face in order to stimulate and facilitate swallowing of saliva or small amounts of food and drink, if considered safe.
  Arms: Intensive F.O.T.T.®
Other: Unspecific Stimulation of face and mouth — The intervention consists of positioning the patient and either washing his face, the hands, or brushing teeth, apply lipbalm, with no specific stimulation or facilitation of swallowing
  Arms: Unspecific stimulation of face and mouth

SUMMARY:
This study is a randomized controlled trial (RCT). Patients after severe acquired brain injury (ABI) were randomised in addition to the individual daily rehabilitation program to intensive Facial Oral Tract Therapy (F.O.T.T.®) (intervention group) or unspecific treatment: washing face, brushing teeth, without facilitating swallowing (control group).

The duration of the intervention period was 15 working days (3 weeks). The intervention in both groups was twice a day.

DETAILED DESCRIPTION:
The F.O.T.T.® approach uses structured tactile input and facilitation techniques in meaningful everyday life context, aiming for improving function in the face and oral tract that is as normal as possible. The goal is maximum participation in daily life. The treatment encourages learning of helpful functional movements or patterns of movement for safe swallowing, protection of airway, oral hygiene, eating, drinking, breathing, voice and articulation.

ELIGIBILITY:
Inclusion Criteria:

* Patients with dysphagia caused by severe ABI

Exclusion Criteria:

* congenital brain damage, psychiatric diagnosis, history of head and neck cancer, agitated behaviour, need for tracheostomy tube

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2014-04 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Change in swallowing frequency of saliva. | Change from baseline frequency of swallowing at three weeks.
  EMBI is a measure device, measuring the number of spontaneous and facilitated swallows by electromyographic and bioimpedance signals.
Change in swallowing quality of saliva (speed of laryngeal elevation) | Change from baseline quality of swallowing at three weeks.
  EMBI is a measure device, measuring the speed of laryngeal elevation during spontaneous and facilitated swallows by electromyographic and bioimpedance signals.
Change in swallowing quality of saliva (Range of movement of laryngeal elevation during swallowing) | Change from baseline quality swallowing at three weeks.
  EMBI is a measure device, measuring the range of movement of laryngeal elevation during spontaneous and facilitated swallows by electromyographic and bioimpedance signals.
Change in swallowing quality of saliva (time of pharyngeal closure during swallowing) | Change from baseline quality of swallowing at three weeks.
  EMBI is a measure device, measuring the time of pharyngeal closure during spontaneous and facilitated swallows by electromyographic and bioimpedance signals.
Change in swallowing quality of saliva (pumping jaw movements before swallowing) | Change from baseline quality of swallowing at three weeks.
  EMBI is a measure device, measuring the pumping jaw movements during spontaneous and facilitated swallows by electromyographic and bioimpedance signals.

SECONDARY OUTCOMES:
Severity of Dysphagia | Baseline and three weeks
  Scored on the Penetration Aspiration Scale (PAS) during Fiberoptic Endoscopic Evaluation of Swallowing
Ability to eat and drink | Baseline and three weeks
  Scored on the Functional Oral Intake Scale (FOIS)

IPD SHARING:
Plan to Share IPD: No